CLINICAL TRIAL: NCT00524056
Title: A Randomized, Double Blind, Placebo-Controlled, Crossover, Proof of Concept Study to Evaluate the Effectiveness and Safety of Carisbamate in the Treatment of Essential Tremor
Brief Title: A Proof of Concept Study of the Effectiveness of Carisbamate in the Treatment of Essential Tremor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR014314; CARISEPY2008
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Essential Tremor, Movement Disorders
Keywords: Essential Tremor; Tremor; Anti-epileptic drug (AED)
MeSH Terms: conditions — Essential Tremor; Movement Disorders; Tremor | interventions — S-2-O-carbamoyl-1-o-chlorophenyl-ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 001 (Experimental): Carisbamate two 100 mg tablets twice per day
  Interventions: Drug: Carisbamate
- 002 (Placebo Comparator): Placebo two placebo tablets twice per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carisbamate — two 100 mg tablets twice per day
  Arms: 001
Drug: Placebo — two placebo tablets twice per day
  Arms: 002

SUMMARY:
The purpose of this study is to evaluate the effectiveness, safety and tolerability of carisbamate treatment for the signs, symptoms, and impairment associated with Essential Tremor (ET) compared to placebo treatment. The secondary objective is to evaluate the effect of carisbamate treatment on indicators of affect and mood in patients who have ET compared to placebo treatment.

DETAILED DESCRIPTION:
The hypothesis of the study is that carisbamate will be effective in the treatment of Essential Tremor compared to placebo as measured by the Fahn-Tolosa-Marin Tremor Rating Scale (TRS). This randomized (study medication assigned by chance) study has 3 Phases: Screening/Washout, Double Blind Treatment (the physician and patient do not know the name of the study medication), and Exit. The Double Blind Treatment Phase has 2 Treatment Periods. Since this is a cross-over study, all subjects who complete the full Double Blind Treatment Phase will have the opportunity to take carisbamate. Carisbamate is administered as 100 mg oral tablets. During Treatment Period 1, patients will take 2 tablets of their assigned study medication (either carisbamate or placebo) two times a day for 21 days. Patients will return for clinical evaluations approximately 1 week after starting the study medication and at the end of Treatment Period 1. Patients will then reduce their dose of study medication to 1 tablet twice a day for 3 days prior to stopping all study medication for at least 11 days. Before entering Treatment Period 2, patients will return for a clinical evaluation. During Treatment Period 2, patients will take 2 tablets of their assigned study medication two times a day for 21 days. Patients will return for clinical evaluations approximately 1 week after starting the second study medication and at the end of Treatment Period 2. Patients will then reduce their study medication to 1 tablet twice a day for 3 days before stopping all study medication. Patients will return for a clinical evaluation approximately 1 week after stopping all study medication and will be contacted by telephone approximately 30 days after the last dose of study medication. Safety will be assessed during each study visit by monitoring adverse events, clinical laboratory testing, physical and neurological examinations and electrocardiograms. Patients will take 2 carisbamate 100mg tablets 2 times a day (400 mg/day) for 21 days during one Treatment Period and 2 matching placebo tablets 2 times a day for 21 days during the other Treatment Period. Patients will reduce the dose of study medication for 3 days at the end of each Treatment Period. There will be times during the study when no study medication is taken.

ELIGIBILITY:
Inclusion Criteria:

* Patients in good general health
* Definite ET based on the TRIG diagnostic criteria
* Patients must have tremor affecting both upper extremities and at least 1 upper extremity must have a postural or action/intention tremor that is rated from 2 (moderate) to 4 (severe) as defined in Part A (Tremor location/severity rating) of the TRS at the Visit 2 evaluation
* Patients must have a negative urine drug screen at screening with exceptions for legally prescribed benzodiazepines or opioid analgesics. Patients must have a negative blood alcohol test at screening and be willing to abstain from alcohol for at least 24 hours prior to each study visit.

Exclusion Criteria:

* Abnormal neurologic signs or progressive neurological disorders, such as Parkinson's Disease, brain tumor, demyelinating disease, CNS trauma, active CNS infection, stroke, or any CNS disease, other than ET, that could interfere with the evaluation of tremor
* Patients with dystonia or dystonic tremors, enhanced physiologic tremor, task specific tremor (e.g., writing tremor), or historical or clinical evidence of psychogenic or fictitious movement disorders
* Patients currently taking or recently exposed to prohibited medications unless, in the opinion of the study investigator, the patient is able to follow the washout procedure and restrictions described in the protocol prior to randomization
* Patients taking more than one tremor-reducing agent who are unable to discontinue all or all but one of these medications
* Patients who have achieved no discernable tremor reduction after treatment with at least 2 of 3 following tremor-reducing medications specifically prescribed for the treatment of ET: propranolol, primidone, or topiramate
* Prior exposure to carisbamate (RWJ-333369)
* Surgical procedures for treatment of ET such as deep brain stimulation or thalamic ablation
* Current or past (within 1 year) major psychotic disorder, such as schizophrenia or other psychotic conditions, major depressive disorder with psychotic features or other psychiatric disorders
* Exacerbation of major depression within the past 6 months
* History of suicide attempts or suicidal ideation in the past year
* History of drug or alcohol abuse within the past year
* Patients who are not able to abstain from alcohol consumption for 24 hours prior to each evaluation
* Patients with abnormal screening laboratory values or ECG (electrical heart tracing)
* Patients with a history, diagnosis or clinical signs for a significant major medical disorder that might disqualify.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-08; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
The primary efficacy outcome is the overall normalized, restricted Tremor Rating Scale (TRS) score after carisbamate treatment compared to placebo treatment. | At baseline, week 1, and week 3 in each treatment period

SECONDARY OUTCOMES:
Overall normalized TRS score; overall normalized unrestricted TRS score, raw TRS total score, raw TRS subscale scores, normalized TRS subscale scores | At baseline, week 1, and week 3 in each treatment period
Profile of Mood States (POMS) | At baseline, then at week 3 in treatment period 1 and at week 3 in treatment period 2
Center for Epidemiological Studies Depression Scale (CES-D) | At baseline, then at week 3 in treatment period 1 and at week 3 in treatment period 2
Rationale for Quality of Life in Essential Tremor questionnaire (QUEST) | At baseline, then at week 3 in treatment period 1 and at week 3 in treatment period 2

CONTACTS AND LOCATIONS:
Overall Officials: Ortho-McNeil Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Ortho-McNeil Janssen Scientific Affairs, LLC

REFERENCES:
- [Derived] Elble RJ, Biondi DM, Ascher S, Wiegand F, Hulihan J. Carisbamate in essential tremor: brief report of a proof of concept study. Mov Disord. 2010 Apr 15;25(5):634-8. doi: 10.1002/mds.22872. PMID 20201005